CLINICAL TRIAL: NCT05825898
Title: Outcome of Patients with Severe Functional Tricuspid Regurgitation
Brief Title: Outcome of Patients with Severe Functional TR According to Medical, Transcatheter or Surgical Treatment
Acronym: TRIGISTRY
Status: Enrolling by invitation | Type: Observational
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, David Messika-Zeitoun, Principal investigator, Ottawa Heart Institute Research Corporation
Other Study IDs: TRIGISTRY
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Conservative management: Patients with TR who did not undergo a tricuspid valve intervention
  Interventions: Procedure: Surgery or Transcatheter tricuspid valve intervention
- Isolated tricuspid valve surgery: Patients with TR who underwent a Isolated tricuspid valve surgery.
  Interventions: Procedure: Surgery or Transcatheter tricuspid valve intervention
- Transcatheter tricuspid valve intervention: Patients with TR who underwent a transcatheter tricuspid valve intervention.
  Interventions: Procedure: Surgery or Transcatheter tricuspid valve intervention

INTERVENTIONS:
Procedure: Surgery or Transcatheter tricuspid valve intervention — Isolated tricuspid valve surgery or Transcatheter tricuspid valve intervention

SUMMARY:
Tricuspid regurgitation (TR) is a public health problem: moderate / severe TR are common, especially in ageing populations, and affect 4% of the population >75 years old, totaling approximately 1.6 million in the US and 3 million in Europe. TR is associated with an increased risk of mortality and morbidity. Contrasting with TR prevalence and the magnitude of the problem, the vast majority of patients are medically treated with diuretics to relieve their symptoms and a curative surgical treatment for isolated severe TR is seldom performed. Reluctance to perform an ITVS can be explained in the one hand by the limited evidence that TR correction improves outcomes and on the other hand, ITVS is associated to high observed in-hospital mortality rates (≈ 10% remarkably consistent in most series across the literature). Severity of the clinical presentation is the main predictor of outcome after surgery. The TRI-SCORE, is a dedicated, simple and accurate risk score model to predict in-hospital mortality after ITVS that could guide the clinical decision-making process at the individual level. Excellent outcomes can be achieved when patients present with low TRI-SCORE. These results suggest adopting a more pro-active approach for TV interventions, and to intervene earlier in the course of the disease in patients with severe isolated TR, irrespective of TR mechanism / etiology, before the occurrence of advanced / irreversible consequences such as severe RV dilatation / dysfunction, renal and liver failure, and intractable heart failure. Recently transcatheter tricuspid valve interventions (TTVI) have emerged recently as a less invasive option to surgery to cure patients with TR.

What is the best treatment between medical, surgical or transcatheter therapy to consider and the best timing for each patient are not clearly defined. The aim of the study is to compare outcome of patients with significant functional TR according to medical, transcatheter or surgical treatment after matching per TRISCORE.

DETAILED DESCRIPTION:
Tricuspid regurgitation (TR) is a public health problem: moderate / severe TR are common, especially in ageing populations, and affect 4% of the population >75 years old, totaling approximately 1.6 million in the US and 3 million in Europe. The literature is consistent showing that TR is a serious condition, associated with morbidity (reduction in exercise capacity, heart failure) and mortality that increase with TR severity.

Current American College of Cardiology (ACC) / American Heart Association (AHA) and European Society of Cardiology (ESC) / European Association of Cardio-Thoracic Surgery guidelines (EACTS) guidelines recommend performing an isolated tricuspid valve surgery (ITVS) in patients with severe secondary (and primary) TR (with or without previous left-sided surgery), who are symptomatic or have right ventricle (RV) dilatation, in the absence of severe RV or left ventricular (LV) dysfunction and severe pulmonary vascular hypertension.

Contrasting with TR prevalence and the magnitude of the problem, the vast majority of patients are medically treated with diuretics to relieve their symptoms and a curative surgical treatment for isolated severe TR is seldom performed ITVS represents only 8% of all tricuspid valve (TV) surgeries and a tricuspid valve intervention is mostly performed at the same time that left-sided heart valve surgery. Thus, only 10% of patients admitted in France with a diagnosis of significant TR are referred for an intervention.

Reluctance to perform an ITVS can be explained in the one hand by the limited evidence that TR correction improves outcomes. Indeed, there is no large randomized multicentric study in the literature to compare medical vs surgical treatment of TR. A recent study did not show difference in long-term survival for patients who undergo surgical intervention compared to medical management alone but this was a non-randomized retrospective single-center study with a small propensity matched sample (62 patients in each group) and matching was performed according to parameters that are not specific to the RV. On the other hand, ITVS is associated to high observed in-hospital mortality rates (≈ 10% remarkably consistent in most series across the literature). In a large French multicentric registry of 466 patients gathering all consecutive patients who underwent a non-congenital ITVS on native valve for severe TR at 12 tertiary centers during a 11-year period (2007-2017), in-hospital mortality was 10% as in other series, but this average rate was hiding important disparities. Mortality rate was indeed markedly variable and was predicted by the severity of the pre-operative clinical, biological and echocardiographic presentation while TR mechanism / etiology had limited impact. As there is no dedicated STS risk score model for ITVS, and the logistic EuroSCORE and the EuroSCORE II were not designed for ITVS, the investigators have developed TRI-SCORE, a dedicated, simple and accurate risk score model to predict in-hospital mortality after ITVS that could guide the clinical decision-making process at the individual level. TRI-SCORE was based on eight clinical (age ≥70 years, NYHA functional class III-IV, right-sided heart failure signs, daily dose of furosemide ≥125 mg), laboratory (glomerular filtration rate <30 ml/min, elevated total bilirubin) and echocardiographic (LV ejection fraction <60%, moderate/severe RV dysfunction) parameters easy to ascertain and capturing the impact of TR on the RV, the liver and the kidneys. This risk score model, on a 0-12 points scale, provided both an excellent discrimination (C-index >0.75) and calibration with a predicted mortality rate ranging from 1% for 0 point to 65% for ≥9 points irrespective of TR mechanism / etiology. Half of patients were referred for an intervention late in the course of the disease with moderately (4-6) or severely elevated (>6) scores, and therefore high mortality rates. In contrast, low in-hospital and 1-year mortality rates (0% to 4%) were achieved in patients with low score (≤3). Our results suggest adopting a more pro-active approach for TV interventions, and to intervene earlier in the course of the disease in patients with severe isolated TR, irrespective of TR mechanism / etiology, before the occurrence of advanced / irreversible consequences such as severe RV dilatation / dysfunction, renal and liver failure, and intractable heart failure.

Transcatheter tricuspid valve interventions (TTVI) are still at an early stage with a large number of percutaneous TV devices currently under development. TTVI are mostly a repair, especially edge-to-edge repair, with promising initial results in the first real world registries with patients at high surgical risk. Therefore, TTVI, as a less-invasive alternative to surgery, may push for an extension of the number of patients treated.

What is the best treatment between medical, surgical or transcatheter therapy to consider and the best timing for each patient are not clearly defined. The aim of the study is to compare outcome of patients with significant functional TR according to medical, transcatheter or surgical treatment after matching per TRISCORE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Isolated (no left-valvular heart disease (mitral regurgitation) >2)
* AND Functional
* AND Moderate to severe or severe Tricuspid regurgitation

Exclusion Criteria:

* Congenital valvular disease,
* Previous tricuspid valve intervention,
* Organic tricuspid valvular disease
* Associated valvular heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enrolled 3 populations of patients with isolated functional TR
  * Patients who remained under conservative management
  * Patients who underwent an isolated valve surgery
  * Patients who underwent a transcatheter valve intervention
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Survival at 2 years | 2 years
  Mortality

SECONDARY OUTCOMES:
Survival free of heart failure admission at 2 years | 2 years
  Patients alive and never admitted for heart failure
Survival and heart failure readmissions | up to 10 years
  Patients alive or never admitted for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: David Messika-Zeitoun, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (44):
- United States (4):
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Health System, New York, New York
- Vienna Medical University, Vienna, Austria
- Canada (4):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - IUCPQ, Québec
  - St Michael's Hospital, Toronto
  - St Paul Hospital, Vancouver
- France (12):
  - Amiens University Hospital, Amiens
  - Henri Mondor Hospital, Créteil
  - CHU Lille, Lille
  - Department of Cardiovascular Surgery and Transplantation, Louis Pradel Cardiovascular Hospital, Lyon
  - APHM, La Timone Hospital, Cardiology Department, Marseille
  - Department of Cardiology, University Hospital of Nancy-Brabois, Nancy
  - CHU de Nantes, Nantes
  - Department of Cardiology, Bichat Claude Bernard Hospital, Paris
  - CHU de RENNES, Rennes
  - CHU Charles Nicolle, Rouen
  - Cardiology Department, Centre Cardiologique du Nord, Saint-Denis
  - Rangueil University Hospital, Toulouse
- Germany (11):
  - Herz- und Diabeteszentrum, Bad Oeynhausen
  - Charité Universitätsmedizin Berlin, Berlin
  - Bonn University Hospital, Bonn
  - University of Cologne, Cologne
  - Cardiovascular center Frankfurt, Frankfurt
  - Albertinen Heart and Vascular Center, Hamburg
  - Asklepios clinic Sankt Georg, Hamburg
  - University Heart and Vascular Center, Hamburg
  - Leipzig University Hospital, Leipzig
  - University Medical Center of Mainz, Mainz
  - Munich Großhadern, Munich
- Tel Aviv Medical center, Tel Aviv, Israel
- Italy (2):
  - Instituto Auxologico Italiano, IRCCS, Milan
  - San Raffaele University Hospital, Milan
- Leiden University Medical center, Leiden, Netherlands
- Spain (5):
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Puerta de Hierro, Madrid
- Switzerland (3):
  - Hopital Universitaire de Bern, Bern
  - Istituto Cardiocentro Ticino, Lugano
  - Zurich Heart Center, Zurich

IPD SHARING:
Plan to Share IPD: No
we have a steering committee which will organize the publication plan